CLINICAL TRIAL: NCT00019825
Title: Phase I Study of Decitabine Mediated Induction of Tumor Antigen and Tumor Suppressor Gene Expression in Lung Cancer Patients
Brief Title: Decitabine in Treating Patients With Unresectable Lung or Esophageal Cancer or Malignant Mesothelioma of the Pleura
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067228; NCI-99-C-0129; NCI-T99-0012; NCT00001824 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2004-07

CONDITIONS: Esophageal Cancer; Lung Cancer; Malignant Mesothelioma; Metastatic Cancer
Keywords: recurrent non-small cell lung cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; advanced malignant mesothelioma; recurrent malignant mesothelioma; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; malignant pleural effusion
MeSH Terms: conditions — Esophageal Neoplasms; Lung Neoplasms; Mesothelioma, Malignant; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Pleural Effusion, Malignant | interventions — Decitabine

INTERVENTIONS:
Drug: decitabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of decitabine in treating patients who have unresectable lung or esophageal cancer or malignant mesothelioma of the pleura.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the pharmacokinetics, toxicity, and maximum tolerated dose of decitabine in patients with unresectable primary small cell or non-small cell lung cancer, unresectable esophageal cancer, or malignant pleural mesothelioma.
* Measure the expression of NY-ESO-1 in tissue samples of these patients before and after receiving this drug.
* Assess the serologic response to NY-ESO-1 in these patients before and after receiving this drug.
* Measure the expression of p16 tumor suppressor gene in these patients before and after receiving this drug.

OUTLINE: This is a dose-escalation study for each stratification group. Patients are stratified according to number of prior therapies (2 or fewer vs 3 or more).

Patients receive decitabine IV continuously on days 1-3. Treatment repeats every 5 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease after completion of the second course receive 2 additional courses.

Cohorts of 3-6 patients receive escalating doses of decitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined for a particular stratum, additional patients from that stratum are treated at the MTD.

Patients are followed for 1 month.

PROJECTED ACCRUAL: A maximum of 72 patients (36 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed unresectable primary small cell lung cancer (SCLC) or non-small cell lung cancer (NSCLC), unresectable esophageal cancer, malignant pleural mesothelioma, or pleural effusions secondary to extrathoracic malignancies
* Disease must be readily accessible to biopsy by endoscopy or percutaneous fine-needle aspiration
* Extrathoracic metastatic disease allowed if no evidence of active intracranial or leptomeningeal metastases

  * Patients treated with prior resection or radiotherapy for intracranial metastatic disease may be eligible provided there is no evidence of active disease on two MRIs (taken one month apart) and patients require no anticonvulsant medications or steroids to control residual symptoms
* No limited stage SCLC or operable NSCLC

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 6 months

Hematopoietic:

* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 10 g/dL
* WBC greater than 3,500/mm^3

Hepatic:

* PT normal
* Bilirubin less than 1.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.6 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* Any of the following conditions require clearance by a cardiologist:

  * Prior coronary artery disease
  * Prior transmural myocardial infarction
  * Congestive heart failure
  * Fixed defects on thallium scan with ejection fraction greater than 40%
* No unstable angina
* No recent deep venous thrombosis requiring anticoagulation

Pulmonary:

* FEV1 and DLCO greater than 30% of predicted
* pCO_2 less than 50 mm Hg
* pO_2 greater than 60 mm Hg on room air
* No recent pulmonary embolism requiring anticoagulation

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 30 days since prior biologic therapy for the malignant tumor

Chemotherapy:

* No prior decitabine
* At least 30 days since other prior chemotherapy for the malignant tumor

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* See Disease Characteristics
* At least 30 days since prior radiotherapy for the malignant tumor (14 days for localized radiotherapy to nontarget lesions) and recovered

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10

CONTACTS AND LOCATIONS:
Overall Officials: David S. Schrump, MD, Study Chair — NCI - Surgery Branch
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Center for Cancer Research, Bethesda, Maryland

REFERENCES:
- [Background] Weiser TS, Guo ZS, Ohnmacht GA, Parkhurst ML, Tong-On P, Marincola FM, Fischette MR, Yu X, Chen GA, Hong JA, Stewart JH, Nguyen DM, Rosenberg SA, Schrump DS. Sequential 5-Aza-2 deoxycytidine-depsipeptide FR901228 treatment induces apoptosis preferentially in cancer cells and facilitates their recognition by cytolytic T lymphocytes specific for NY-ESO-1. J Immunother. 2001 Mar-Apr;24(2):151-61. doi: 10.1097/00002371-200103000-00010. PMID 11265773
- [Background] Weiser TS, Ohnmacht GA, Guo ZS, Fischette MR, Chen GA, Hong JA, Nguyen DM, Schrump DS. Induction of MAGE-3 expression in lung and esophageal cancer cells. Ann Thorac Surg. 2001 Jan;71(1):295-301; discussion 301-2. doi: 10.1016/s0003-4975(00)02421-8. PMID 11216765